CLINICAL TRIAL: NCT03267823
Title: Comparison of INR Determined by Point-of-Care to Standard Laboratory Testing Before and After Reversal of Heparin in Cardiac Surgery
Brief Title: INR Comparison Testing in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Michael Fabbro, Assistant Professor, University of Miami
Other Study IDs: 20170003
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Coagulation Disorder
Keywords: Bleeding; heart surgery; coagulation; coagulopathy; INR
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart surgery: Patients undergoing heart surgery will have blood samples tested for INR values
  Interventions: Diagnostic Test: International Normal Ratio (INR)

INTERVENTIONS:
Diagnostic Test: International Normal Ratio (INR) — Blood test for INR using laboratory and point of care methods

SUMMARY:
The investigator is testing blood samples to compare the results of two different techniques. Since blood loss and the need for blood transfusions continue to be major problems after heart surgery and other types of surgery, the blood clotting levels are constantly checked during heart surgery as part of clinical care.The purpose of this study is to compare the INR levels in blood before and after the heart bypass during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age.
* Patients undergoing elective surgery.
* Patients undergoing cardiac surgery.
* Patients to undergo general anesthesia with endotracheal intubation.
* Patients with well-controlled health disorders.

Exclusion Criteria:

* Patients currently on Coumadin or other anticoagulants; including, direct thrombin inhibitors and direct Xa inhibitors.
* Patients who are under 18 years of age or pregnant.
* Patients undergoing emergency surgery.
* Patients with known coagulation disorders.
* Patients who are unable to provide informed consent in the form of a signature

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Change in correlation between laboratory and point of care INR | Baseline, Within ten minutes of completion of bypass
  Pearson's Coefficient

SECONDARY OUTCOMES:
Change in agreement between laboratory and point of care INR | Baseline, Within ten minutes of completion of bypass
  Bland-Altman plots

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fabbro, DO, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fabbro M 2nd, Abalo M, Fermin L, Andrews DM, Patel PA. Comparison of international normalized ratio determined by point-of-care to standard laboratory testing before and after reversal of heparin in cardiac surgery. Blood Coagul Fibrinolysis. 2020 Mar;31(2):140-144. doi: 10.1097/MBC.0000000000000889. PMID 31934886